CLINICAL TRIAL: NCT01905072
Title: Preventing Childhood Obesity Through Early Feeding and Parenting Guidance
Brief Title: Preventing Childhood Obesity Through Early Guidance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arizona State University (Other)
Responsible Party: Principal Investigator, Elizabeth Reifsnider, Associate Dean of Research, Arizona State University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 1R01DK096488-01A1 (NIH); GRANT11114271 (Other: Arizona State University)
Record Dates: First submitted 2013-07-16; First posted 2013-07-23 (Estimated); Last update posted 2020-01-18 (Actual); Status verified 2020-01

CONDITIONS: Childhood Obesity
Keywords: Obesity; Breastfeeding; Educational Intervention
MeSH Terms: conditions — Pediatric Obesity; Obesity; Breast Feeding

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Education Home Visits (Experimental): The intervention group will receive the full intervention delivered by community health workers (CHWs) through home visits. CHWs will deliver the intervention in the subjects' homes. Home visits will be arranged at subjects' convenience and occur on a planned schedule. The intervention content will be based on the Institute of Medicine recommendations.
  Interventions: Other: Education Home Visits
- Control Group (No Intervention): The control group will receive only measurement visits, with no intervention or interaction during the home visits. They will receive only support from their WIC clinic.

INTERVENTIONS:
Other: Education Home Visits — Intervention will include educational home visits on:
  1. Growth monitoring and feedback
  2. Feeding: support exclusive breastfeeding until 6 months; delay solid feeding until 6 months; appropriate amounts of food for age; stop bottle feeding at 12 months; have nothing but breast milk/formula/4 oz juice in bottle; limit juice amount to 4 oz day; introduce cup by 10-11 months; no sweetened beverages; limited amounts of sweets.
  3. Parenting: recognizing hunger and satiety cues; handling colic/crying; engaging baby in play.
  4. Activity: being active with the baby; no screen time for baby and limited to 1 hour for 1-3 year olds; promote active play while maintaining safety.
  5. Sleep: at least 10-12 hours sleep per day needed; how to promote sleeping environment for baby.
  Arms: Education Home Visits

SUMMARY:
The goal of this study is to compare the effectiveness of structured CHW- provided home visits, using an intervention created through community-based participatory research, to standard care received through WIC office visits in preventing the development of overweight (weight/length >85th percentile) and obesity (weight/length >95th percentile) in infants during their first 2 years of life.

Hypothesis 1: Children in the intervention group will remain within their growth centiles in height/weight and weight for age, while children in the control group will increase in height/weight percentiles and weight percentiles more rapidly (> .67 SD) during the first year of life.

Hypothesis 2: Fewer children who receive the intervention will have BMI >95th percentile at ages 2 and 3 than the children in the control group.

Hypothesis 3: Children who receive the intervention will exclusively breastfeed for a longer period of time than will children in the control group.

Hypothesis 4: Children who receive the intervention will have a higher percentage of fruits and vegetables and a lower percentage of sweetened beverages, desserts, and candy in their diets at ages 1, 2, and 3, than will children in the control group.

Hypothesis 5: Parents in the intervention group will be more responsive to infant feeding cues (hunger, satiety)than parents in the control group.

DETAILED DESCRIPTION:
Along with birth weight and parental body size, infant feeding is recognized as one of the most influential biological and environmental factors that affect weight gain during infancy. Parental feeding practices have a strong impact on children's food availability, eating behaviors, and weight. The Institute of Medicine's(IOM) recent report (2011) on early childhood obesity prevention policies recommends five approaches to preventing obesity: assess, monitor, and track growth from birth to age 5; increase physical activity and decrease sedentary behavior in young children; support breastfeeding and be responsive to children's feeding cues; limit screen time; and promote age-appropriate sleep for young children. Based on the previous work by this research team, and in collaboration with a major urban health department, we propose to test an intervention that incorporates all the IOM's recommendations to prevent the development of obesity in at-risk infants. The intervention will be guided by health professionals and delivered through home visits by community health workers (CHWs), supervised by public health nurses (PHN), to Mexican American women and children who are clients of the Special Supplemental Nutrition Program for Women, Infants, and Children (WIC) Program in Houston, TX. The intervention will occur for 2 years with 1 year of follow-up, for a total of 3 years of measures.

ELIGIBILITY:
Inclusion Criteria:

MATERNAL - Self-described as Mexican American, pre-pregnant BMI of 25 or greater, speaks English or Spanish, is between the ages of 18 and 40, lives in a home where she can receive home visitors, has no diagnosed chronic diseases that can affect the growth of a fetus (cardiac, respiratory, etc.), have a telephone contact, and is not intending to move from the area. Gestational diabetes will be noted but is not an exclusion criterion; however, Type 1 diabetics will be excluded. Exposure to tobacco smoke (either maternal or household smoking) will be noted as it is associated with infant obesity, but will not be an inclusion or exclusion criteria.

INFANT - We will enroll the full-term singleton infants of enrolled mothers. The infants will be enrolled if they are > 38 weeks gestation, have a birth weight > 2500 gm, and are without endocrine/chromosomal/genetic abnormality that could interfere with growth.

Exclusion Criteria:

MATERNAL - Not enrolled in WIC clinic or does not plan to continue with WIC clinic after delivery, high-risk pregnancy, hospitalized after discharge of infant, separated from infant, or experiencing significant postpartum complications. If these criteria develop in an enrolled mother, she will remain in the study per CONSORT guidelines, but her infant will not be followed for study outcomes. We have sufficient power with our sample size to allow for these events.

INFANT - Not discharged home with the mother or who are otherwise separated from their mothers or who has a severe illness that can affect growth. CONSORT guidelines will apply in these cases as well as in maternal cases.

Ages: 1 Day to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 177 (Actual)
Dates: Start 2012-10; Primary Completion 2017-06-30 (Actual); Study Completion 2017-06-30 (Actual)

PRIMARY OUTCOMES:
Weight for Length Body Mass Index | BMI will be assessed at three years of age for the study participants
  The children in the study will be compared at age three (intervention and control group) for differences in weight, height, and Body Mass index.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth A Reifsnider, PhD RN FAAN, Principal Investigator — Arizona State University
Locations (1):
- St. Austin Center - Arizona State University Group, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: Yes
We will make our data available through our website. All data will be de-identified and will not be able to be altered but can be downloaded (with permission from PI) for secondary analysis.

REFERENCES:
- [Derived] Reifsnider E, McCormick DP, Cullen KW, Szalacha L, Moramarco MW, Diaz A, Reyna L. A randomized controlled trial to prevent childhood obesity through early childhood feeding and parenting guidance: rationale and design of study. BMC Public Health. 2013 Sep 24;13:880. doi: 10.1186/1471-2458-13-880. PMID 24063435